CLINICAL TRIAL: NCT06716515
Title: Influence of Gender Difference on Knee Proprioception in Non-Specific Low Back Pain Among Young Adults
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norhan Yousif Allam, Teaching Assistant, Cairo University
Other Study IDs: P.T.REC/012/005429
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Non-Specific Chronic Low-back Pain
Keywords: Gender Difference; Knee Proprioception; Chronic Non-Specific Low-back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males: Forty-one males will be evaluated using digital inclinometer in an open kinetic chain position. The JPS testing is conducted in the sitting position without feet floor contact, at a quiet place with closed eyes . Investigator will perform all the knee joint position sense assessments in the dominant extremity. The digital inclinometer is stabilized to the middle third of the subjects' leg (15 cm distal from the apex of the fibular head) with a strap. The starting position of the test is 90° flexion. The proprioception evaluation angle is defined at 30°. Participants are asked to extend their tested knee to the target angle of 30° from the initial position (90° knee flexion) then to return to their initial position after 5 seconds in this position ,The participant indicated by saying "YES" when they thought they reach the target, and the reposition accuracy will be measured as the joint position error (JPE) in degrees, as displayed on the digital inclinometer screen
  Interventions: Device: digital inclinometer
- Females: Forty-one females will be assessed the same as group A , Then compare Results To investigate the impact of gender difference on knee proprioception among non specific low back pain young adults
  Interventions: Device: digital inclinometer

INTERVENTIONS:
Device: digital inclinometer — Digital inclinometer to assess gender difference in knee repositioning error

SUMMARY:
the aim of the study is to investigate the impact of gender difference on knee proprioception among non specific low back pain young adults.

DETAILED DESCRIPTION:
Low back pain (LBP) is one of the most common musculoskeletal disorders and the leading causes of disability and work absence globally. LBP notonly causes individual suffering, but also a heavy burden to the society. Despite this, up to 85% patients with LBP cannot be clearly diagnosed and are classified as non-specific LBP (NSLBP). Proprioception plays an important role in the planning of precise and coordinated movements, in maintaining balance and controlling body posture. It also exerts its influence on motor learning and re-education. Proprioception deficit has been identified in people with LBP and it has been suggested that these deficits might be associated with causes and mechanisms of LBP. Although the local investigation of proprioception is important, the proprioceptive deficits due to LBP may not be restricted only to the lumbar region. Anatomical and biomechanical associations between the knee and lower back segments imply that the knee might be adversely affected in patients with LBP.

there is a gap in the literature concerning sex differences in the knee joint proprioception. Although biomechanical and hormonal differences between males and females are suspected to be responsible for increasing this incidence.

ELIGIBILITY:
Inclusion Criteria:

1. Forty-one Patients from each gender participated in the study.
2. Subject's age ranged from 18-26 years old, with Body Mass Index (BMI) less than 30Kg/m2
3. The dominant knees of the subjects (defined as the leg used for kicking) are tested.
4. Pain between three and eight using numerical pain rating scale NPRS, and Oswestry Disability Index score less than 20.
5. All the subjects sign an informed consent form. 6. able to comprehend and follow the examiner's instructions.

Exclusion Criteria:

1. limitation of active and passive knee joint motion.
2. clinical signs of an impairment or abnormality in the knee (such as abnormal range of motion, muscle weakness, or malalignment).
3. injury to the knee that required medical attention.
4. current pain in the knee or previous surgery on the knee.
5. not able to understand and follow the commands of the examiner.

Ages: 18 Years to 26 Years | Sex: All
Age Groups: Adult
Study Population: Eighty-two Young Adults (include males and females), ranging in age from 18 to 26, will be included in the study. Individuals will be assigned into 2 groups. Group (A) 41 males with non specific low back pain (B) 41 females with non specific low back pain.
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
knee proprioception | up to 4 weeks
  knee repositioning error is measured by digital inclinometer

SECONDARY OUTCOMES:
Functional disability | up to 4 weeks
  measured by Oswestry disability index (arabic version)

OTHER OUTCOMES:
Pain intensity | up to 4 weeks
  measured by Numerical rating scale( each subject choose a number from 0 to 10)